CLINICAL TRIAL: NCT06252974
Title: Accurate Diagnosis of the Invasion Depth in Early Esophageal Squamous Cell Carcinoma by a Deep Neural Network Analysis of Narrow-band Imaging Endoscopy Data
Brief Title: Accurate Diagnosis of the Invasion Depth in ESCC by a Deep Neural Network Analysis of NBI Endoscopy Data
Status: Not yet recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LY2023-229-B
Record Dates: First submitted 2024-01-22; First posted 2024-02-12 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to accurate diagnose the stage of esophageal squamous cell carcinoma in order to help physicians to decide the appropriate clinical treatment. The main question it aims to answer is:

• To get early accurate diagnosis of the invasion depth of esophageal squamous cell carcinoma by narrow-band imaging endoscopy data.

Participants' clinical informations from routine examinations and treatments will be collected, there will be no harm to participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, regardless of gender;
2. Performing esophageal ESD surgery due to esophageal mucosal lesions;
3. Pathological evaluation of ESD specimens.

Exclusion Criteria:

Pathological examination after ESD surgery ruled out esophageal squamous cell carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Around 500 cases.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04-25 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Accurate diagnose the invasion depth of early esophageal squamous cell carcinoma by endoscopy NBI images through deep neural network analysis | 2024/12/31
  We will compare the predictive performance of InvaDepNet before and after incorporating data generated using GAN and demonstrated that including the generated data in the training dataset effectively improves the accuracy of the predictive model. Additionally, we will train six commonly used CNN models on two datasets with different shooting angles (including NBI without magnifying and NBI with magnifying), and we will propose a ResNet model to analysis the clinical informations combine with NBI images.